CLINICAL TRIAL: NCT01103934
Title: The Addition of Vitamin D to Fluticasone Propionate in the Management of Seasonal Allergic Rhinitis
Brief Title: Vitamin D Plus Fluticasone Propionate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-184-B
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Cholecalciferol; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Propionate plus Vitamin D3 (Active Comparator): Subjects will be treated with fluticasone propionate and Vitamin D once daily for 2 weeks during allergy season
  Interventions: Drug: Vitamin D3; Drug: Fluticasone Propionate
- Fluticasone Propionate plus Placebo (Placebo Comparator): Subjects will be treated with fluticasone propionate and placebo for Vitamin D once daily for 2 weeks during allergy season
  Interventions: Drug: Placebo; Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Vitamin D3 — 4000 IU once daily
  Arms: Fluticasone Propionate plus Vitamin D3
Drug: Placebo — Placebo taken once daily
  Arms: Fluticasone Propionate plus Placebo
Drug: Fluticasone Propionate — 200 mcg daily, intranasal
  Other Names: Flonase

SUMMARY:
The objectives of this study would be to see if the addition of vitamin D to fluticasone propionate provides greater symptomatic relief in patients with seasonal allergic rhinitis compared to fluticasone propionate treatment alone.

ELIGIBILITY:
Inclusion Criteria

1. Males and females between 18 and 45 years of age.
2. History of tree, grass and/or ragweed allergic rhinitis.
3. Positive skin test to tree, grass and/or ragweed antigen.
4. Positive response to screening nasal challenge.

Exclusion Criteria

1. Physical signs or symptoms suggestive of renal, hepatic or cardiovascular disease.
2. Pregnant or lactating women.
3. Upper respiratory infection within 14 days of study start.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Naclerio, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluticasone Propionate Plus Vitamin D3 | Fluticasone Propionate Plus Placebo
Started | 17 | 18
Completed | 17 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate Plus Vitamin D3 | Fluticasone Propionate Plus Placebo | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (6.1) | 29.5 (9.3) | 28.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Nasal Symptom Score (TNSS) Over 2 Week Randomized Treatment Period
Description: Patients recorded the severity of sneezing, runny nose, stuffy nose, and other symptoms (e.g. itchy nose/throat) twice a day on a scale from 0 to 3 (0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe). The TNSS was calculated as the sum of all scores for morning and evening recordings with a range of 0 to 24. The change from baseline for each day of treatment was then calculated for each subject. So that each subject only had one observation, the average of these changes was calculated for each subject, and this summary measure was used in the analysis comparing the two treatment groups. We report the median and full range of these average changes for each group. A negative value indicates an improvement in symptoms.
Time Frame: Baseline and 2 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fluticasone Propionate Plus Vitamin D3 | Fluticasone Propionate Plus Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | -11.3 [-18.9 to 8.8] | -7.6 [-18.7 to 0.7]
Statistical Analysis 1: Comparison: Fluticasone Propionate Plus Vitamin D3 vs Fluticasone Propionate Plus Placebo; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change From Baseline in Daytime Nasal Symptom Score (DNSS) Over 2 Week Randomized Treatment Period
Description: Patients recorded the severity of sneezing, runny nose, stuffy nose, and other symptoms (e.g. itchy nose/throat) twice a day on a scale from 0 to 3 (0 = no symptoms, 1 = mild, 2 = moderate, and 3 = severe). The DNSS was calculated as the sum of all scores for morning with a range of 0 to 12. The change from baseline for each day of treatment was then calculated for each subject. So that each subject only had one observation, the average of these changes was calculated for each subject, and this summary measure was used in the analysis comparing the two treatment groups. We report the median and full range of these average changes for each group. A negative value indicates an improvement in daytime symptoms.
Time Frame: Baseline and 2 weeks
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Fluticasone Propionate Plus Vitamin D3 | Fluticasone Propionate Plus Placebo
Number analyzed (Participants) | 17 | 18
units on a scale | -6.9 [-10.2 to 5.2] | -3.7 [-10.6 to -0.2]
Statistical Analysis 1: Comparison: Fluticasone Propionate Plus Vitamin D3 vs Fluticasone Propionate Plus Placebo; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Fluticasone Propionate Plus Vitamin D3 | Fluticasone Propionate Plus Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 0/17 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes